CLINICAL TRIAL: NCT03682523
Title: The Breaking "Bad Rest" Study: Interrupting Sedentary Time to Reverse Frailty Levels in Acute Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Olga Theou (Other)
Responsible Party: Sponsor-Investigator, Olga Theou, PhD, Assistant Professor, Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Breaking Bad Rest
Record Dates: First submitted 2018-09-12; First posted 2018-09-24 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Sedentary Lifestyle
Keywords: Frailty; Hospitalization; Acute care; older adults; intervention
MeSH Terms: conditions — Sedentary Behavior; Frailty

STUDY DESIGN:
Intervention Model Description: Participants will be classified into three strata based on their baseline mobility measured with the HABAM. Within each strata, patients will be randomly allocated to the control (n=25) and intervention (n=25) groups in temporal blocks. In the event of Covid-19 related interruptions to the study, temporal blocks aim to keep the number of participants in the intervention and control groups similar at all times.
  This stratified, block randomised control trial design will ensure a similar distribution of patient characteristics in the control and intervention groups and will safeguard against possible interruptions due to Covid-19.
Who Masked: Investigator, Outcomes Assessor
Masking Description: A senior statistician will use a computer-generated random sequence to determine whether each patient is allocated to the control or intervention group. To minimize risk of bias, the RA who collects assessment data will remain blinded to the study group, with separate RAs assisting with the intervention. Only the statistician will hold the key to the control/intervention group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Fitted with an accelerometer to measure time spent out of bed while in hospital. Otherwise, participants in the control group will receive usual care from the hospital medical team during their hospital stay. Daily activities of participants will not be restricted if patients are assigned to the control group.
- Intervention Group (Experimental): Fitted with accelerometer to measure time spent out of bed while in hospital; daily goals set for time spent out of bed; mobilization feedback real-time feedback on goal attainment; hands on mobilization by physiotherapist for participants in late afternoon for participants who do not meet daily goal.
  Interventions: Behavioral: Sedentary behavior reduction intervention

INTERVENTIONS:
Behavioral: Sedentary behavior reduction intervention — Participants will be provided with a device to measure physical activity and sedentary behaviours. A tablet will be in the research office and each afternoon, it will be synced to the device to assess the activity progress of the patient. The research team will deliver an upright time goal and will target a 20% increase in upright time from the previous hospital day. Physiotherapist research assistants will visit the participants every afternoon to monitor progress and safely mobilize participants to their maximum ability if they have not met their daily goal (including weekend). The maximum level of ability will be determined in consultation with the healthcare team. Participants who do not meet their goal will be mobilized in the late afternoon/ early evening.
  Arms: Intervention Group

SUMMARY:
This study will determine whether an intervention aimed at reducing sedentary time in patients admitted to acute care will result in decreased frailty levels at hospital discharge, compared to the current standard of care. All patients will be fitted with accelerometers then randomised to the control or intervention group. The control group will receive only standard of care while in hospital. Participants in the intervention group will engage in daily goal setting for time out-of-bed and have access to real-time feedback on a bedside monitor. Participants in the intervention group will also received assisted mobilization if they have not met their daily goal by the late afternoon. The main outcome is frailty, assessed by a frailty index.

DETAILED DESCRIPTION:
The objective of this study is to determine if an intervention designed to reduce sedentary time during a patient's stay in acute care will reduce patient's frailty levels more so than current standard of care. This study will be conducted at a single-centre, but will be a stratified, block randomised control trial. Fifty participants will be recruited within 24 hours of admission to a geriatric acute care unit. Both groups will be fitted with a device that measures sedentary and active time (accelerometer). Participants in the intervention group will have a daily goal for activity and will be provided with real-time feedback on attainment of that goal displayed on a bedside tablet. Participants in the intervention group who do not independently achieve their goal will be assisted in reducing their sedentary time in the afternoon and/or early evening to the maximum level of their ability; this level will be determined in consultation with the healthcare team. The primary outcome is a change in frailty during hospitalization, measured using a 30-item frailty index. The data collection phase is approximately 10 months. Data analysis will take an additional six months (16 months total). Knowledge-users will be involved during all stages of the project. The data generated from this study will enable us to scale up this intervention nationally and internationally. If the intervention is successful, it will warrant a study to implement the intervention as part of standard care. Ultimately, this study will inform guidelines to limit patients' sedentary behaviors in acute care.

ELIGIBILITY:
Inclusion Criteria:

* Anticipated hospital length of stay >1 day
* Patient or care partner able to communicate in English

Exclusion Criteria:

* Patient unable to provide informed consent and care partner not available to provide consent
* Bedridden prior to hospital admission
* Previous participation in our study (i.e. readmission during data collection phase)
* End-of-life or waiting for long-term care facility
* Patient is admitted to a shared room with a current study participant.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-04-07 (Actual); Primary Completion 2023-07-20 (Actual); Study Completion 2023-07-20 (Actual)

PRIMARY OUTCOMES:
Change in the Frailty Index | Change from baseline frailty up to a median 14 day hospital length of stay
  The frailty index (FI) operationalizes frailty in clinical practice and for research. FI scores are calculated as the proportion of potential deficits present in a given individual. For this study we will construct a 30-item FI using a health questionnaire administered to patients or their care partners (if patients are not able to self-report) at each study time point. The proportion of patients changing their FI scores by >=0.1 from baseline to hospital discharge is the primary outcome.
  Data collection is opportunistic, based on length of stay. The discharge date is not fixed - thus day-in-study at discharge will not be the same for all participants. Depending on length of stay, participants will provide data for additional time points between baseline and discharge, including week 1, week 2, week 3, week 4 and then in 30 day intervals. However, not every participant will have the same number of time points. Note that the median hospital length of stay is 14 days.

SECONDARY OUTCOMES:
Change in the Frailty Index | Change from baseline frailty up to a median 14 days hospital length of stay, and 30 days after hospital discharge
  The frailty index (FI) operationalizes frailty in clinical practice and for research. FI scores are calculated as the proportion of potential deficits present in a given individual. For this study we will construct a 30-item FI using a health questionnaire administered to patients or their care partners (if patients are not able to self-report) at each study time point. Secondary outcome for the FI is a change from baseline up to one month following hospital discharge as a continuous measure.
  Data collection is opportunistic, based on length of stay. The discharge date is not fixed - thus day-in-study at discharge will not be the same for all participants. Depending on length of stay, participants will provide data for additional time points between baseline and discharge, including week 1, week 2, week 3, week 4 and then in 30 day intervals. However, not every participant will have the same number of time points. Note that the median hospital length of stay is 14 days.
Change in upright time | Change from baseline upright time up to a median 14 day hospital length of stay
  Time (minutes/day) spent upright out of bed (upright time) will be tracked continuously during the participants' hospital length of stay using accelerometers for both groups. Patients will be fitted with accelerometers within 24 hours of admission. An ActivatorTM (PAL Technologies Ltd) accelerometer will be attached to the mid-thigh of the patients' dominant side.
  Data collection is opportunistic, based on length of stay. The discharge date is not fixed - thus day-in-study at discharge will not be the same for all participants. Depending on length of stay, participants will provide data for additional time points between baseline and discharge, including week 1, week 2, week 3, week 4 and then in 30 day intervals. However, not every participant will have the same number of time points. Note that the median hospital length of stay is 14 days.
Change in upright bouts | Change from baseline upright bouts up to a median 14 day hospital length of stay
  The number of times/day that a participants gets upright out of bed (upright bouts) will be tracked continuously during the participants' hospital length of stay using accelerometers for both groups. Patients will be fitted with accelerometers within 24 hours of admission. An ActivatorTM (PAL Technologies Ltd) accelerometer will be attached to the mid-thigh of the patients' dominant side.
  Data collection is opportunistic, based on length of stay. The discharge date is not fixed - thus day-in-study at discharge will not be the same for all participants. Depending on length of stay, participants will provide data for additional time points between baseline and discharge, including week 1, week 2, week 3, week 4 and then in 30 day intervals. However, not every participant will have the same number of time points. Note that the median hospital length of stay is 14 days.
Change in mobility: Hierarchical Assessment of Balance and Mobility (HABAM) | Change from baseline mobility scores up to a median 14 day hospital length of stay
  The HABAM is a clinical tool used to obtain a global measure of a patients' health through the assessment of mobility, transfers and balance. Patients receive daily scores based on demonstrated ability in each focal area; testing if the patient can move around in bed, sit up in bed, stand up, etc. The median hospital length of stay is expected to be 14 days, but many patients will have a longer length of stay. This means that some patients will have more data collection time points than others.
Change in balance: Hierarchical Assessment of Balance and Mobility (HABAM) | Change from baseline balance scores up to a median 14 day hospital length of stay
  The HABAM is a clinical tool used to obtain a global measure of a patients' health through the assessment of mobility, transfers and balance. Patients receive daily scores based on demonstrated ability in each focal area; testing if the patient can move around in bed, sit up in bed, stand up, etc. The median hospital length of stay is expected to be 14 days, but many patients will have a longer length of stay. This means that some patients will have more data collection time points than others.
Falls | From baseline to 30 days after hospital discharge
  The number of falls will be assessed by reviewing medical charts during hospitalization and by self-report at the one month follow-up.
Hospital length of stay | From baseline up to a median 14 day hospital length of stay
  Medical chart reviews will be assessed to measure hospital length of stay
In-hospital mortality | From baseline up to a median 14 day hospital length of stay
  Medical chart reviews will be assessed to measure in-hospital mortality
Hospital readmissions | From baseline up to 30 days after hospital discharge
  Medical chart reviews will be assessed to measure readmissions within 30 days.
Safety evaluation (frequency of adverse events) | From baseline up to a median 14 day hospital length of stay
  Safety will be determined through medical chart audit for frequency of adverse events
Cost | From baseline up to 30 days after hospital discharge
  Costs (Canadian Dollars) related to the interventions will be collected prospectively from the intervention accounts and costs incurred by the healthcare system and patients will be collected through interviews and follow-up surveys, respectively. An appropriate decision-analytic modeling framework will be employed to undertake cost-effectiveness analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Olga Theou, PhD, Principal Investigator — Assistant Professor, Department of Medicine, Dalhousie University
Locations (1):
- QEII Health Sciences Centre, Halifax, Nova Scotia, Canada

REFERENCES:
- [Background] Hoogerduijn JG, Buurman BM, Korevaar JC, Grobbee DE, de Rooij SE, Schuurmans MJ. The prediction of functional decline in older hospitalised patients. Age Ageing. 2012 May;41(3):381-7. doi: 10.1093/ageing/afs015. Epub 2012 Feb 28. PMID 22378613
- [Background] Covinsky KE, Palmer RM, Fortinsky RH, Counsell SR, Stewart AL, Kresevic D, Burant CJ, Landefeld CS. Loss of independence in activities of daily living in older adults hospitalized with medical illnesses: increased vulnerability with age. J Am Geriatr Soc. 2003 Apr;51(4):451-8. doi: 10.1046/j.1532-5415.2003.51152.x. PMID 12657063
- [Background] Chong E, Ho E, Baldevarona-Llego J, Chan M, Wu L, Tay L. Frailty and Risk of Adverse Outcomes in Hospitalized Older Adults: A Comparison of Different Frailty Measures. J Am Med Dir Assoc. 2017 Jul 1;18(7):638.e7-638.e11. doi: 10.1016/j.jamda.2017.04.011. Epub 2017 Jun 3. PMID 28587850
- [Background] Romero-Ortuno R, Forsyth DR, Wilson KJ, Cameron E, Wallis S, Biram R, Keevil V. The Association of Geriatric Syndromes with Hospital Outcomes. J Hosp Med. 2017 Feb;12(2):83-89. doi: 10.12788/jhm.2685. PMID 28182802
- [Background] Romero-Ortuno R, Wallis S, Biram R, Keevil V. Clinical frailty adds to acute illness severity in predicting mortality in hospitalized older adults: An observational study. Eur J Intern Med. 2016 Nov;35:24-34. doi: 10.1016/j.ejim.2016.08.033. Epub 2016 Sep 2. PMID 27596721
- [Background] Baldwin C, van Kessel G, Phillips A, Johnston K. Accelerometry Shows Inpatients With Acute Medical or Surgical Conditions Spend Little Time Upright and Are Highly Sedentary: Systematic Review. Phys Ther. 2017 Nov 1;97(11):1044-1065. doi: 10.1093/ptj/pzx076. PMID 29077906
- [Background] Kortebein P, Ferrando A, Lombeida J, Wolfe R, Evans WJ. Effect of 10 days of bed rest on skeletal muscle in healthy older adults. JAMA. 2007 Apr 25;297(16):1772-4. doi: 10.1001/jama.297.16.1772-b. No abstract available. PMID 17456818
- [Background] Lipnicki DM, Gunga HC. Physical inactivity and cognitive functioning: results from bed rest studies. Eur J Appl Physiol. 2009 Jan;105(1):27-35. doi: 10.1007/s00421-008-0869-5. Epub 2008 Sep 17. PMID 18797919
- [Background] Kortebein P, Symons TB, Ferrando A, Paddon-Jones D, Ronsen O, Protas E, Conger S, Lombeida J, Wolfe R, Evans WJ. Functional impact of 10 days of bed rest in healthy older adults. J Gerontol A Biol Sci Med Sci. 2008 Oct;63(10):1076-81. doi: 10.1093/gerona/63.10.1076. PMID 18948558
- [Background] Aguilar-Farias N, Brown WJ, Peeters GM. ActiGraph GT3X+ cut-points for identifying sedentary behaviour in older adults in free-living environments. J Sci Med Sport. 2014 May;17(3):293-9. doi: 10.1016/j.jsams.2013.07.002. Epub 2013 Aug 8. PMID 23932934
- [Background] Egerton T, Brauer SG, Cresswell AG. Fatigue after physical activity in healthy and balance-impaired elderly. J Aging Phys Act. 2009 Jan;17(1):89-105. doi: 10.1123/japa.17.1.89. PMID 19299841
- [Background] Tremblay MS, Carson V, Chaput JP, Connor Gorber S, Dinh T, Duggan M, Faulkner G, Gray CE, Gruber R, Janson K, Janssen I, Katzmarzyk PT, Kho ME, Latimer-Cheung AE, LeBlanc C, Okely AD, Olds T, Pate RR, Phillips A, Poitras VJ, Rodenburg S, Sampson M, Saunders TJ, Stone JA, Stratton G, Weiss SK, Zehr L. Canadian 24-Hour Movement Guidelines for Children and Youth: An Integration of Physical Activity, Sedentary Behaviour, and Sleep. Appl Physiol Nutr Metab. 2016 Jun;41(6 Suppl 3):S311-27. doi: 10.1139/apnm-2016-0151. PMID 27306437
- [Background] Shadmi E, Zisberg A. In-hospital mobility and length of stay. Arch Intern Med. 2011 Jul 25;171(14):1298; author reply 1298-9. doi: 10.1001/archinternmed.2011.321. No abstract available. PMID 21788551
- [Background] Brown CJ, Williams BR, Woodby LL, Davis LL, Allman RM. Barriers to mobility during hospitalization from the perspectives of older patients and their nurses and physicians. J Hosp Med. 2007 Sep;2(5):305-13. doi: 10.1002/jhm.209. PMID 17935241
- [Background] Liu B, Moore JE, Almaawiy U, Chan WH, Khan S, Ewusie J, Hamid JS, Straus SE; MOVE ON Collaboration. Outcomes of Mobilisation of Vulnerable Elders in Ontario (MOVE ON): a multisite interrupted time series evaluation of an implementation intervention to increase patient mobilisation. Age Ageing. 2018 Jan 1;47(1):112-119. doi: 10.1093/ageing/afx128. PMID 28985310
- [Background] Hartley PJ, Keevil VL, Alushi L, Charles RL, Conroy EB, Costello PM, Dixon B, Dolinska-Grzybek AM, Vajda D, Romero-Ortuno R. Earlier Physical Therapy Input Is Associated With a Reduced Length of Hospital Stay and Reduced Care Needs on Discharge in Frail Older Inpatients: An Observational Study. J Geriatr Phys Ther. 2019 Apr/Jun;42(2):E7-E14. doi: 10.1519/JPT.0000000000000134. PMID 28628498
- [Background] Hartley P, Adamson J, Cunningham C, Embleton G, Romero-Ortuno R. Higher Physiotherapy Frequency Is Associated with Shorter Length of Stay and Greater Functional Recovery in Hospitalized Frail Older Adults: A Retrospective Observational Study. J Frailty Aging. 2016;5(2):121-5. doi: 10.14283/jfa.2016.95. PMID 27224504
- [Background] Eklund K, Wilhelmson K, Gustafsson H, Landahl S, Dahlin-Ivanoff S. One-year outcome of frailty indicators and activities of daily living following the randomised controlled trial: "Continuum of care for frail older people". BMC Geriatr. 2013 Jul 22;13:76. doi: 10.1186/1471-2318-13-76. PMID 23875866
- [Background] Mitnitski AB, Mogilner AJ, Rockwood K. Accumulation of deficits as a proxy measure of aging. ScientificWorldJournal. 2001 Aug 8;1:323-36. doi: 10.1100/tsw.2001.58. PMID 12806071
- [Background] de Vries NM, Staal JB, van Ravensberg CD, Hobbelen JS, Olde Rikkert MG, Nijhuis-van der Sanden MW. Outcome instruments to measure frailty: a systematic review. Ageing Res Rev. 2011 Jan;10(1):104-14. doi: 10.1016/j.arr.2010.09.001. Epub 2010 Sep 17. PMID 20850567
- [Background] Theou O, O'Connell MD, King-Kallimanis BL, O'Halloran AM, Rockwood K, Kenny RA. Measuring frailty using self-report and test-based health measures. Age Ageing. 2015 May;44(3):471-7. doi: 10.1093/ageing/afv010. Epub 2015 Feb 16. PMID 25687601
- [Background] Hubbard RE, Peel NM, Samanta M, Gray LC, Mitnitski A, Rockwood K. Frailty status at admission to hospital predicts multiple adverse outcomes. Age Ageing. 2017 Sep 1;46(5):801-806. doi: 10.1093/ageing/afx081. PMID 28531254
- [Background] Laporte M, Keller HH, Payette H, Allard JP, Duerksen DR, Bernier P, Jeejeebhoy K, Gramlich L, Davidson B, Vesnaver E, Teterina A. Validity and reliability of the new Canadian Nutrition Screening Tool in the 'real-world' hospital setting. Eur J Clin Nutr. 2015 May;69(5):558-64. doi: 10.1038/ejcn.2014.270. Epub 2014 Dec 17. PMID 25514899
- [Background] Lord S, Chastin SF, McInnes L, Little L, Briggs P, Rochester L. Exploring patterns of daily physical and sedentary behaviour in community-dwelling older adults. Age Ageing. 2011 Mar;40(2):205-10. doi: 10.1093/ageing/afq166. Epub 2011 Jan 14. PMID 21239410
- [Background] Cowie A, Thow MK, Granat MH, Mitchell SL. A comparison of home and hospital-based exercise training in heart failure: immediate and long-term effects upon physical activity level. Eur J Cardiovasc Prev Rehabil. 2011 Apr;18(2):158-66. doi: 10.1177/1741826710389389. Epub 2011 Feb 18. PMID 21450662
- [Background] Chan CS, Slaughter SE, Jones CA, Ickert C, Wagg AS. Measuring Activity Performance of Older Adults Using the activPAL: A Rapid Review. Healthcare (Basel). 2017 Dec 13;5(4):94. doi: 10.3390/healthcare5040094. PMID 29236062
- [Background] Hubbard RE, Eeles EM, Rockwood MR, Fallah N, Ross E, Mitnitski A, Rockwood K. Assessing balance and mobility to track illness and recovery in older inpatients. J Gen Intern Med. 2011 Dec;26(12):1471-8. doi: 10.1007/s11606-011-1821-7. Epub 2011 Aug 16. PMID 21845488
- [Result] Theou O, Stathokostas L, Roland KP, Jakobi JM, Patterson C, Vandervoort AA, Jones GR. The effectiveness of exercise interventions for the management of frailty: a systematic review. J Aging Res. 2011 Apr 4;2011:569194. doi: 10.4061/2011/569194. PMID 21584244
- [Derived] Theou O, O'Brien MW, Godin J, Blanchard C, Cahill L, Hajizadeh M, Hartley P, Jarrett P, Kehler DS, Romero-Ortuno R, Visvanathan R, Rockwood K. Interrupting bedtime to reverse frailty levels in acute care: a study protocol for the Breaking Bad Rest randomized controlled trial. BMC Geriatr. 2023 Aug 10;23(1):482. doi: 10.1186/s12877-023-04172-x. PMID 37563553